CLINICAL TRIAL: NCT06570395
Title: Osteopathic Manipulative Treatment in the Third Trimester of Pregnancy
Status: Terminated | Type: Observational
Why Stopped: Staff turnover led to difficulty in recruiting.
Sponsor: Corewell Health South (Other)
Responsible Party: Sponsor
Other Study IDs: MMMC#1637
Record Dates: First submitted 2024-08-03; First posted 2024-08-26 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Osteopathic Manipulative Treatment (OMT)
Keywords: Pregnancy; Osteopathic Manipulative Treatment (OMT); Delivery Outcomes; Third Trimester Pregnancy
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OMT Intervention: The OMT intervention group will be patients who consent to participating in OMT through the Southwest Women's Clinic and Cass Community Clinic in Niles, MI.
  Case Inclusion:
  1. Pregnant patients, ages 18-34
  2. Primiparous and multiparous
  3. Gestational age ≥34 weeks
  4. Delivering at Corewell Health South Saint Joseph or Niles hospitals
  5. Consent for treatment or as a control
  Case Exclusion:
  1. Absolute contraindications to OMT
  2. Acute abdomen
  3. BP >160/110
  4. Unexplained visual disturbances
  5. Heavy vaginal bleeding preceding delivery
  6. <34 weeks gestational age
  7. Treatment refusal
  8. Magnesium sulfate received for seizure prophylaxis in setting of preeclampsia w/ severe features or severe gestational HTN
  9. Scheduled c-section due to prior OB conditions
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Control Group: The control group will be patients who consent to participating in the control group through the Southwest Women's Clinic and Cass Community Clinic in Niles, MI.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Osteopathic Manipulative Therapy (OMT) is a hands-on approach to treating conditions that affect all areas of the body. Physicians trained in OMT (Doctors of Osteopathic Medicine or DO) use OMT to correct structural imbalances in the body, relieve pain, and improve circulation. It is not only used as a treatment modality, but also to diagnose and prevent disease and improve overall functioning. There are over 40 OMT techniques that all involve gentle manipulation of the muscles, soft tissues, and joints in several ways to optimize alignment, improve blood flow, restore balance, and improve range of motion ("Osteopathic Manipulative Therapy & OMT." Cleveland Clinic).
  Groups: OMT Intervention

SUMMARY:
Osteopathic Manipulative Therapy (OMT) is a hands-on approach to treating conditions that affect all areas of the body. Physicians trained in OMT (Doctors of Osteopathic Medicine or DO) use OMT to correct structural imbalances in the body, relieve pain, and improve circulation. Research shows that manual therapy is equally or more effective in treating pain and improving function versus oral analgesics (Bodine). OMT can decrease cost and improve function in patients with a minimal adverse effect profile. OMT applications include relieving asthma, irritable bowel syndrome, fibromyalgia, migraines, carpal tunnel syndrome, and sports-related injuries. In addition to the indications listed above, there is a growing body of research surrounding the use of OMT in pregnancy and its use in treatment and prevention of complications peripartum.

Research Question: Does OMT during the third trimester of pregnancy improve delivery outcomes including: decreased labor times, less utilization of analgesics, fewer incidences of meconium fluid and perineal lacerations, and reduced risk of conversion to c-section or operative vaginal delivery? Though all research has shown that OMT is safe in pregnancy, there has been conflicting data on its benefits during the peripartum period. Additional research is needed to show its utility in decreasing labor times and need for analgesics during labor and reducing incidence of adverse outcomes including perineal lacerations and conversion to c-section and operative vaginal delivery. The current study will add to the growing body of knowledge about OMT during pregnancy and its potential benefits outside of musculoskeletal pain relief.

DETAILED DESCRIPTION:
Osteopathic Manipulative Therapy (OMT) is a hands-on approach to treating conditions that affect all areas of the body. Physicians trained in OMT (Doctors of Osteopathic Medicine or DO) use OMT to correct structural imbalances in the body, relieve pain, and improve circulation. It is not only used as a treatment modality, but also to diagnose and prevent disease and improve overall functioning. There are over 40 OMT techniques that all involve gentle manipulation of the muscles, soft tissues, and joints in several ways to optimize alignment, improve blood flow, restore balance, and improve range of motion ("Osteopathic Manipulative Therapy & OMT." Cleveland Clinic). Research shows that manual therapy is equally or more effective in treating pain and improving function versus oral analgesics (Bodine). OMT can decrease cost and improve function in patients with a minimal adverse effect profile.

Some OMT techniques are similar to those used by chiropractors, physical therapists, and massage therapists. What makes it unique is that osteopathic physicians are trained to apply the philosophies of OMT with their comprehensive medical training of all body systems to specifically adapt the treatment to each individual patient. They incorporate their vast knowledge of pathology and physiology with the philosophy that the body can self-heal and self-regulate.

While OMT is most known for its application in treating pain, it truly involves holistic examination of the whole patient - body, mind, and spirit - and can be applied to any situation that places stress upon the body. It is also adjusted based on the patient's condition, age, weight, and other characteristics to yield personalized treatment that can be an adjunct to treatment for virtually any disease or condition (Roberts). Other OMT applications include relieving asthma, irritable bowel syndrome, fibromyalgia, migraines, carpal tunnel syndrome, and sports-related injuries. In addition to the indications listed above, there is a growing body of research surrounding the use of OMT in pregnancy and its use in treatment and prevention of complications peripartum.

The current practice of obstetrics does not often incorporate the use of OMT in pregnancy to treat pain or prevent complications during and after delivery, despite evidence that it is safe. The investigators believe there is a need to focus attention on the effect of OMT on the rates of specific adverse events in labor and delivery.

Research Question: Does OMT during the third trimester of pregnancy improve delivery outcomes including: decreased labor times, less utilization of analgesics, fewer incidences of meconium fluid and perineal lacerations, and reduced risk of conversion to c-section or operative vaginal delivery? Though all research has shown that OMT is safe in pregnancy there has been conflicting data on its benefits during the peripartum period. Additional research is needed to show its utility in decreasing labor times and need for analgesics during labor and reducing incidence of adverse outcomes including perineal lacerations and conversion to c-section and operative vaginal delivery. The current study will add to the growing body of knowledge about OMT during pregnancy and its potential benefits outside of musculoskeletal pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients, ages 18-34
* Primiparous and multiparous
* Gestational age ≥34 weeks
* Delivering at Corewell Health South Saint Joseph or Niles hospitals
* Consent for treatment or as a control

Exclusion Criteria:

* Absolute contraindications to OMT
* Acute abdomen
* BP >160/110
* Unexplained visual disturbances
* Heavy vaginal bleeding preceding delivery
* <34 weeks gestational age
* Treatment refusal
* Magnesium sulfate received for seizure prophylaxis in setting of preeclampsia w/ severe features or severe gestational HTN
* Scheduled c-section due to prior OB conditions

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Patients must be in third trimester of pregnancy to participate.
Study Population: Patients in the third trimester of pregnancy who opt into OMT treatments and meet the inclusion/exclusion criteria of the study.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2024-07-16 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Labor duration | Upon delivery
  Does OMT in the 3rd trimester of pregnancy shorten duration of labor? The investigators will compare a control group to a group who received OMT.

SECONDARY OUTCOMES:
Number of patients with analgesic use during labor | Upon delivery
  Does OMT in the 3rd trimester of pregnancy reduce the use of analgesic during labor? The investigators will compare a control group to a group who received OMT.
Degree of perineal laceration during labor | Upon delivery
  Does OMT in the 3rd trimester of pregnancy reduce the extent of perineal laceration during labor? The investigators will compare a control group to a group who received OMT.
Number of patients with meconium fluid upon delivery | Upon delivery
  Does OMT in the 3rd trimester of pregnancy reduce the presence of meconium fluid upon delivery? The investigators will compare a control group to a group who received OMT.
Number of patients who underwent operative vaginal delivery | Upon delivery
  Does OMT in the 3rd trimester of pregnancy reduce number of patients who undergo operative vaginal delivery? The investigators will compare a control group to a group who received OMT.
Number of patients who were converted to c-section | Upon delivery
  Does OMT in the 3rd trimester of pregnancy reduce number of patients who converted to C-section during delivery? The investigators will compare a control group to a group who received OMT.

CONTACTS AND LOCATIONS:
Overall Officials: Max Schaefer, DO, Principal Investigator — Corewell Health South
Locations (1):
- Corewell Health Lakeland, Saint Joseph, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carnes D, Mars TS, Mullinger B, Froud R, Underwood M. Adverse events and manual therapy: a systematic review. Man Ther. 2010 Aug;15(4):355-63. doi: 10.1016/j.math.2009.12.006. Epub 2010 Jan 22. PMID 20097115
- [Background] Roberts A, Harris K, Outen B, Bukvic A, Smith B, Schultz A, Bergman S, Mondal D. Osteopathic Manipulative Medicine: A Brief Review of the Hands-On Treatment Approaches and Their Therapeutic Uses. Medicines (Basel). 2022 Apr 27;9(5):33. doi: 10.3390/medicines9050033. PMID 35622072
- [Background] Bodine WA. Osteopathic Manipulative Treatment: A Primary Care Approach. Am Fam Physician. 2019 Feb 15;99(4):214. No abstract available. PMID 30763051

DOCUMENTS (1):
  • Study Protocol (2025-05-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT06570395/Prot_000.pdf